CLINICAL TRIAL: NCT05058417
Title: Assessment of Empagliflozin as Adjuvant Therapy in Patients With Ulcerative Colitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Institutional and funding constrains
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Principle Investigator, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G12/2021
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin group (Experimental): participants will receive 10 mg Empagliflozin for 8 consecutive weeks in addition to the standard therapy
  Interventions: Drug: Empagliflozin 10 MG
- Placebo (Placebo Comparator): participants will receive placebo for 8 consecutive weeks in addition to the standard therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — participants will receive 10 mg Empagliflozin for 8 consecutive weeks in addition to the standard therapy
  Arms: Empagliflozin group
Drug: Placebo — participants will receive placebo for 8 consecutive weeks in addition to the standard therapy
  Arms: Placebo

SUMMARY:
This is a randomized, controlled study evaluating empagliflozin tablets administered daily for 8 weeks. The purpose of the study is to evaluate the efficacy and safety of empagliflozin in the treatment of mild to moderately active ulcerative colitis. Disease activity will be measured using Mayo score for ulcerative colitis activity. Calculation of the score requires patients to undergo colonoscopy at the start of the study and at week 8.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild or moderate ulcerative colitis newly diagnosed by colonoscopy and biopsy according to Mayo endoscopic scoring of ulcerative colitis.
* Adults (males and/or females) with age range from 18 to 65 years old.
* Patients on treatment with 5-aminosalisylic acid (5-ASA)

Exclusion Criteria:

* Patients with severe ulcerative colitis according to Mayo endoscopic scoring of ulcerative colitis.
* Treatment with systemic or rectal steroids.
* Treatment with immunosuppressants.
* Previously failed treatment with a sulphasalazine.
* Known hypersensitivity to any of study drugs.
* Hepatic and renal dysfunction.
* Pregnancy and lactation.
* History of colorectal carcinoma.
* History of complete or partial colectomy.
* Patients with diabetes mellitus
* Patients with history of lactic acidosis
* Patients with disease states associated with hypoxemia including cardiorespiratory insufficiency
* Positive stool culture for enteric pathogens, positive stool ova and parasite exam.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Expression of colonic (NF)-κB proteins | 8 weeks
  Difference between the two groups in the expression of colonic (NF)-κB proteins.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF